CLINICAL TRIAL: NCT04370132
Title: Segment IV Hypertrophy After Liver Venous Deprivation Compared to Portal Embolization in Patient Before Major Hepatectomy
Brief Title: Segment IV Hypertrophy After Liver Venous Deprivation
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0212
Record Dates: First submitted 2020-04-17; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Major Hepatectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group of patient with liver venous deprivation: Group of patient with liver venous deprivation
- Group of patient with portal embolization: Group of patient with portal embolization

SUMMARY:
before major hepatectomy, in case of insufisant future liver remanent volume or function, portal embolization is a routinely used method to enable growth of the future liver remnant. Recently liver venous deprivation has been described in some pioneer centre. The results are processing with greater and faster hypertrophy allowing probably less drop out from the embolization to surgery compared to portal embolization.

In major hepatectomy, and specially in right or extended right hepatectomy the segment IV plays an important role in the proportion of future liver remnant.

Despite the growing interest in the scientific community for liver venous deprivation many aspects concerning the liver hypertrophy remains unexplored. In particular the the degree of hypertrophy of segment IV after liver venous deprivation compared to portal embolization.

ELIGIBILITY:
Inclusion criteria:

- patient with liver tumor selected for right hepatectomy with insufficient future liver remnant who have undergoes portal embolization or liver venous deprivation

Exclusion criteria:

- left / extended left hepatectomy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with liver tumors selected for surgery with insufficient futur liver remnant
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
segment IV degree of hypertrophy | 1 day
  segment IV degree of hypertrophy

SECONDARY OUTCOMES:
overall survival | 5 years
  overall Survival : overall survival : is overall survival from date of hepatic surgery until the 01/04/2020 or during 5 years
recurrence free survival | 5 years
  recurrence free Survival : is the the survival without same deasese recurrence from the hepatic surgery date until the 01/04/2020 or during 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio PANARO, PhD, Study Director — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC